CLINICAL TRIAL: NCT03323073
Title: Study of Functional Networks in Resting fMRI as Biomarkers of Monopolar or Bipolar Depression
Brief Title: Study of Functional Networks in Resting fMRI
Acronym: DEPIMAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Deadline of the end date of the inclusions
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: FoundaMental Mental Health Foundation RTRS (France) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P100144
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Acute Depression; Major Depressive Episode
Keywords: unipolar; bipolar; depression; resting state fMRI; neural network; connectivity
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bipolar disorder type I or II (Active Comparator): a single resting state fMR for patients with bipolar disorder type I or II with acute depressive state
  Interventions: Other: Resting state fMRI
- Unipolar disorder (Active Comparator): a single resting state fMR for patients with monopolar disorder with acute depressive state
  Interventions: Other: Resting state fMRI
- Healthy volunteers (Other): a single resting state fMRI for subjects without psychiatric disorders assessed by the SCID
  Interventions: Other: Resting state fMRI

INTERVENTIONS:
Other: Resting state fMRI — One single fMRI which is used to characterize a uni or a bipolar major depressive episode (MDE).

SUMMARY:
The primary purpose is to compare with resting fMRI the functional networks of rest (RTS) in unipolar depression and in bipolar depression.

Hypothesis : the main objective of this work is to compare with the rest fMRI the Rest Functional Networks (RFN) in the unipolar depression and in the bipolar depression in order to identify specific biomarkers for each affection. The general hypothesis of this work is that intra- and inter RFN connectivity is different between bipolar patients and unipolar patients. Specifically the investigators assume that connectivity within the default mode network (including ventral mediofrontal cortex, subgenual cingulate cortex, inferior parietal cortex, posterior cingulate cortex) will be increased in unipolar patients compared to bipolar patients.

DETAILED DESCRIPTION:
Study hypothesis:

The investigators assume that connectivity within the DMR will be increased in unipolar patients compared to bipolar patients. Similarly the investigators assume, in agreement with the results of our studies using N-Back (Harvey et al, 2005) and studies in self reference process in the unipolar depression (Grimm et al, 2009; and Lemogne al, 2009) that the DMR and frontoparietal networks connectivity (intraparietal cortex and dorsolateral prefrontal cortex) will be unusually positive in unipolar patients compared to bipolar patients.

Methods:

Transversal, multicenter, comparative study evaluating unipolar and bipolar patients in depressive phase and controls group without psychiatric disorders. The study involves one single assessment with fMRI, which is used to characterize a mono or bipolar major MDE. The question is not to predict subsequent progression towards a unipolar or bipolar disorder.

Primary outcome :

Comparison of unipolar and bipolar depressed patients in depressive acute phase and control subjects with fMRI resting task and an itself reference task and a diffusion tensor sequence. Patients will be evaluated clinically by: the MADRS, the YMRS, the BDRS, the Mathys, the SCID.

Secondary outcome:

verifying the RFR functional integrity in bipolar depression or unipolar by comparing the brain activity patterns of depressed patients than the control group;

Experimental arm: patient with bipolar disorder type I or II and patient with unipolar disorder Control arm: subjects without psychiatric disorders assessed by the SCID Number of patients per arm : 40 Total number of patients : 123 Duration : inclusions 3 years. Duration of inclusion per patient : 16 days Number of participating centres : 4 Statistical analyses: fMRI data analysis strategy

The primary criterion is the variation of BOLD signal during resting state and during self-referential processing task in both groups of depressed patients compared to control group. Functional connectivity within and between DMN (default mode network), CEN (central executive network) and SN (salience network) will be tested using a multivariate approach, independent component analysis (ICA). This analysis simultaneously decomposes group fMRI data into modes describing variations across space, time per subject to identify independent functional spatial maps corresponding to coherent brain functional networks.

A between-group analysis of variance (ANOVA) will be performed to assess the difference of functional connectivity within and between DMN, CEN and SN comprising a between factor group (unipolar, bipolar, controls) for resting state data and data from the self-referential task.

Correlations:

Correlations will be explored between fMRI parameters (in default mode and central executive network) and clinical criteria (e.g scores in MATTIS, MADRSn, YMRS).

ELIGIBILITY:
Inclusion Criteria:

* Unipolar and bipolar depressed patients including patients with type I and type II bipolar disorders.
* Patients in an acute depressive state (according to DSM-IV criteria).
* Men or Women with age between 18 to 65 years.
* Patients with unipolar depression must fullfill Mitchel's criteria for unipolar depression.
* MADRS score > 22
* YMRS score < 12
* Mean duration of depressive episode < 1 year
* in-patient or out-patient

Healthy volunteers matched for age and socio-educational level, without personal history of unipolar or bipolar depression and without psychiatric disorders

Exclusion Criteria:

Patients and controls:

* Bipolar disorder with rapid cycling
* Suicidal thoughts with score > 3 at the MADRS item 'suicide'
* Depression with psychotic features
* Psychiatric co-morbidity including other AXIS-1 disorders (OCD, schizophrenia, social phobia) and borderline personality disorder
* Substance and alcohol abuse or dependance
* Recent treatment with ECT (< 6 months)
* Previous history of Brain Traumatic Injury; neurological disorders (multiple sclerosis, parkinson's disease, stroke) or disorders associated with abnormal MRI (lupus, Behcet's disease)
* Contra-indication of MRI: pregnancy; tatoos; claustrophobia
* Patient hospitalized under legal condition
* Patient that requires an important sedation due to anxiety
* Bipolar patients that requires at less 3 mood stabilizers
* Patient receiving a new antidepressant since more than 10 days
* Patients without social security insurance
* Patients with legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2014-11-18 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Bold signal and connectivity coefficients within and between neural networks | one day (within 16 days after inclusion)
  Bold connectivity assessed with resting state fMRI within and between networks

SECONDARY OUTCOMES:
Correlations between clinical scores (MADRS, YMRS, SCID) and neural network connectivity. | one day (within 16 days after inclusion)
  Relationship between clinical variables and scores of connectivity within and between networks in unipolar and bipolar depressed patients
Sensibility and specificity of fMRI to predict unipolar and bipolar depressive status | one day (within 16 days after inclusion)
  relationships between clinical variables and scores of connectivity within and between networks in unipolar and bipolar depressed patients

CONTACTS AND LOCATIONS:
Overall Officials: Philippe FOSSATI, Professor, Principal Investigator — AP-HP, Pitié-Salpêtrière Hospital of Paris

IPD SHARING:
Plan to Share IPD: No